CLINICAL TRIAL: NCT00892450
Title: Anticholinergic Therapy for Overactive Bladder in Parkinson's Disease: A Randomized, Double-blind, Crossover Pilot Study
Brief Title: Anticholinergic Therapy for Overactive Bladder in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 01143
Record Dates: First submitted 2009-04-28; First posted 2009-05-04 (Estimated); Last update posted 2014-10-03 (Estimated); Status verified 2014-10

CONDITIONS: Parkinson's Disease; Overactive Bladder
Keywords: Overactive bladder symptoms; Parkinson's disease; darifenacin; oxybutynin; cognition
MeSH Terms: conditions — Parkinson Disease; Urinary Bladder, Overactive | interventions — oxybutynin; darifenacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental): crossover design
  Interventions: Drug: Oxybutynin and darifenacin

INTERVENTIONS:
Drug: Oxybutynin and darifenacin — Participants with overactive bladder will take each medication for 4 weeks.

SUMMARY:
The purpose of this research study is to investigate the cognitive (thinking, memory, knowledge, intelligence) side effects of two medications commonly used to treat overactive bladder (OAB) symptoms in veteran patients with Parkinson's disease (PD) seen at the Philadelphia PADRECC.

DETAILED DESCRIPTION:
This study will be a double-blinded cross-over clinical trial design to assess the prevalence of cognitive effects, the efficacy, and the effect on quality of life (QOL) of two anticholinergic medications commonly used in the treatment of overactive bladder (OAB): oxybutynin and darifenacin. This will be done by use of a well-established and validated computer-based cognitive battery. Secondary endpoints will assess efficacy of anticholinergic therapy on symptoms of OAB via QOL questionnaire and participant urinary diaries.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic PD (ICD9=332.0)
* MMSE 24, able to give informed consent and complete questionnaires and voiding diaries.
* Urological work-up within 3 months of enrollment to:

  * Rule out treatable causes of urinary symptoms

    * Urinalysis (UA)
    * Post-void residual ultrasound (PVR)
    * Urinary cytology
  * Documented symptoms OAB on screening 3-day voiding diary:

    * Average of 1 urgency episode / 24 hours, and
    * Average of 8 micturitions / 24 hours
    * Subjective complaints of symptoms for 3 months

Exclusion Criteria:

* Exposure to anticholinergics or antispasmodics within the last 4 weeks (among them: atropine, tolterodine, benztropine, trihexyphenidyl, dicyclomine, hyoscyamine, and scopolamine)
* Exposure to drugs with known effects on cognition (i.e. opioids, benzodiazepines or sedating antihistamines) within the last week
* Exposure to drugs contraindicated or cautioned in use with the 2 study medications (drugs that also use the cytochrome P450 enzyme, primarily CYP3A4). These include: ketoconazole, itraconazole, miconazole, erythromycin, clarithromycin, ritonavir, nelfinavir, nefazodone, flecainide, thioridazine and tricyclic antidepressants.
* Nonpharmacological treatment of OAB within the last 4 weeks (for example: biofeedback, physical therapy, acupuncture)
* Uncontrolled narrow angle glaucoma
* History of gastric or urinary retention / dysmotility (ulcerative colitis, myasthenia gravis and severe constipation)
* History of hepatic or renal impairment
* History of severe gastro-esophageal reflux disease and/or use of bisphosphonates, patients at risk for esophagitis
* Previous exposure to anticholinergic for OAB symptoms that resulted in side effects that caused cessation of the medication

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-05; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
compare cognitive side effects | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jayne R Wilkinson, MD, Principal Investigator — VA Medical Center, Philadelphia
Locations (1):
- VA Medical Center, Philadelphia, Philadelphia, Pennsylvania, United States